CLINICAL TRIAL: NCT04385615
Title: Effect of Fasting Mimicking Diet on the Activation of Beige/Brown Adipose Tissue in Humans
Brief Title: Fasting Mimicking Diet and Beige/Brown Adipose Tissue in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Marcela Reymond Simoes, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAAE: 20037719.0.0000.5404
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Obesity
Keywords: Obesity; Fasting Mimicking Diet (FMD); Brown Adipose Tissue (BAT)
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: One group will receive the FMD diet. The other group will be the control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMD Group (Experimental): Participants will be requested to follow a Fasting Mimicking Diet, for three consecutive months. Before and after the intervention dietary intake and physical activity data, evaluation of beige/brown adipose tissue activation, anthropometric measures and body composition (DEXA scan), lipid profile and inflammatory markers.
  Interventions: Other: Fasting Mimicking Diet
- Control Group (No Intervention): Participants will be requested to continue with their habitual eating habits, for three consecutive months. Before and after the intervention dietary intake and physical activity data, evaluation of beige/brown adipose tissue activation, anthropometric measures and body composition (DEXA scan), lipid profile and inflammatory markers.

INTERVENTIONS:
Other: Fasting Mimicking Diet — Participants will be requested to follow three cycles (of 5 day each), for three consecutive months, of a Fasting Mimicking Diet, a plant-based, low-calorie, low-protein, low-carbohydrate, high-unsaturated fat diet. For the remaining 25 days of each month, participants should continue with their habitual eating habits.
  Arms: FMD Group

SUMMARY:
Obesity today has become one of the main public health concerns. As a consequence, different strategies have arisen to fight weight gain. One of the alternative strategies to increase the success of therapeutic approaches to weight loss is the increase in energy expenditure, through thermogenesis, regulated by the beige/brown adipose tissue (BAT). Studies have shown that beige/BAT has a strong correlation with body weight regulation. It has also been demonstrated that cold exposure activates beige/BAT. Recent studies, mainly in animal models, suggest that beige/BAT can also be activated by specific food and nutrients. Concomitantly, new dietary interventions, to treat obesity, have also been studied. One of these dietary interventions is the Fasting Mimicking Diet (FMD). Since FMD is high in unsaturated fat, and clinical trials have shown that FMD interventions reduced body weight and improved metabolic health, there is a possible association between this diet and the activation of beige/BAT. The aim of this is study is to investigate the effect of Fasting Mimicking Diet on the activation of beige/brown adipose tissue, in humans with overweight. This will be an open clinical trial with the duration of three consecutive months (three cycles of the FMD diet). There will be an FMD and a control group. The following data will be collected before and after the intervention, for each group: dietary intake and physical activity data, evaluation of beige/brown adipose tissue activation (Positron Emission Tomography - PET with fluoride-18-labeled fluorodeoxyglucose (18F-FDG) in combination with computed tomography - PET/CT scan, Thermal Imaging, BAT adipokines and genes related to BAT activity), basal metabolic rates and caloric needs (Indirect Calorimetry), anthropometric measures and body composition (DEXA scan), lipid profile and inflammatory markers. Data will be expressed as mean and standard deviation and the variables will be compared by Student's t-test or ANOVA, for repeated measures.

DETAILED DESCRIPTION:
HYPOTHESIS

Beige/BAT has been shown as a promising strategy to treat obesity. The exact mechanism, and stimulus, of activation of this tissue have not been completely clarified. However, some studies have identified some nutrients, such as unsaturated fat, as a potential stimulus for activation. The effect of Fasting Mimicking Diet on the activation of Beige/Brown Adipose Tissue has not yet been investigated. Since FMD is high in unsaturated fat, and clinical trials have shown that FMD interventions reduced body weight and improved metabolic health, there is a possible association between this diet and the activation of beige/BAT.

Our hypothesis is that an intervention, with a 5-days cycle for 3 consecutive months, of Fasting Mimicking Diet will promote beige/brown adipose tissue activation and will improve body weight and metabolic markers related to obesity, in humans with overweight.

OBJECTIVES

Main Objective

To evaluate the effect of a dietary intervention using 3 cycles of Fasting Mimicking Diet on the activation of beige/brown adipose tissue, in humans with overweight.

Specific Objectives

* To evaluate the effect of the FMD on the activation of Beige/Brown Adipose Tissue using PET/CT (FDG-18) and Thermal Imaging (FLIR camera);
* To evaluate anthropometric measures (weight, abdomen circumference) and body composition (DEXA scan), before, during and after the FMD intervention;
* To evaluate basal metabolic rates and daily caloric needs (Indirect Calorimetry), before and after the FMD intervention;
* To evaluate the effect of the FMD on metabolic markers and hormones: leptin (ELISA), insulin (ELISA), glucose, total cholesterol, LDL, HDL and triglycerides;
* To evaluate the effect of the FMD on insulin sensitivity (using OGIS);
* To evaluate the effect of the FMD on cytokines: tumor necrosis factor alpha (TNF-α), interleukin 1-beta (IL1β), Monocyte Chemoattractant Protein-1 (MCP1), interleukin-6 (IL-6) and interleukin-10 (IL-10) (ELISA);
* To evaluate the effect of the FMD on Brown Adipose Tissue Adipokines: insulin-like growth factor 1 (IGF-1), IL-6, fibroblast growth factor 21 (FGF21) and 12,13-dihydroxy-9z-octadecenoic acid (12,13-diHOME) (ELISA);
* To evaluate the effect of the FMD on BAT activation genes: peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α) and G-protein coupled receptor 120 (GPR120) (PCR).

MATERIALS AND METHODS

Selection of Participants

The estimated sample size is 26 individuals. Participants will be overweight. There will be a control group (n=13) and an FMD group (n=13). There will be similar sample size for both genders. Participants will be recruited through electronic and printed media propagation.

Design

This will be an open clinical trial with the duration of three consecutive months (three cycles). There will be data collection before, during and after the dietary intervention. In this intervention, participants will be requested either to follow three cycles of a Fasting Mimicking Diet, or to follow their habitual eating habits for three months (control group). For the FMD group, participants will receive the FMD diet and will be requested to follow the recommendations from the manufacturer: FMD diet for 5 consecutive days (during these days, they will be asked to only eat the FMD diet), and for the remaining 25 days of the month, participants should continue with their habitual eating habits. This procedure will be repeated three times.

The FMD diet will be provided by L-Nutra, Nutrition for Longevity (commercial name of the diet: ProLon). All the data will be collected at University of Campinas, Brazil. More specifically, the Indirect Calorimetry and the DEXA scan will be done at the LIMED (Laboratory of Investigation of Metabolism and Diabetes) and the PET/CT (FDG-18) will be done at the Center of Nuclear Medicine in the Hospital de Clínicas (HC) Hospital.

The following data will be collected from both groups (control and FMD):

* Evaluation of food consumption: 24hr-Food Recall - before, during and after the intervention;
* Evaluation of physical activity: short version of the International Physical Activity Questionnaire IPAQ) - before and after the intervention;
* Evaluation of beige/BAT activity:

  * Positron Emission Tomography (PET) with fluoride-18-labeled fluorodeoxyglucose (18F-FDG) in combination with computed tomography (PET/CT scan) - before and after the intervention:
  * Individualized cooling protocol: For this exam, participants will be allocated in a room with a controlled temperature (19oC). They will be using light cloths and a cooling vest (commercial name: Polar), for one hour. Right after, they will receive 4.0 megabecquerel/kg (MBq/kg) of 18F-FDG and will continue in the room, with a controlled temperature (19oC), for another hour. After these two hours they will move to the PET/CT room;
  * Thermal Imaging (FLIR camera) - before, during and after the intervention:
  * Individualized cooling protocol: For this exam, participants will be allocated in a room with a controlled temperature (19oC). They will be using light cloths and a cooling vest (commercial name: Polar), for two hours;
  * Brown Adipose Tissue Adipokines: IGF-1, IL-6, FGF21 and 12,13-diHOME, using ELISA;
  * Brown Adipose Tissue activation genes: PGC-1α and GPR120, using PCR;
* Evaluation of basal metabolic rates and caloric needs: Indirect Calorimetry (gas exchange analysis: oxygen (O2) consumption and carbon dioxide (CO2) release) - before and after the intervention;
* Evaluation of anthropometric measures - before, during and after the intervention:

  * Weight (digital scale) and height (fixed stadiometer);
  * Abdominal circumference;
  * Body composition: Dual-energy X-ray absorptiometry (DEXA scan);
* Blood samples - before, during and after the intervention:

  * Cytokines (TNF-α, IL1β, MCP1, IL-6 and IL-10) and hormones (insulin and leptin) - Enzyme-linked immunosorbent assay (ELISA);
  * Metabolic markers (glucose, total cholesterol, LDL, HDL and triglycerides);
  * Insulin sensitivity - OGIS (Oral Glucose Insulin Sensitivity). This measurement is calculated using insulin and glucose values.

Statistical Analysis

Data will be expressed as mean and standard deviation and the variables will be compared by Student's t-test or ANOVA, for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 25 and < 30kg/m2.

Exclusion Criteria:

* Residing outside of Campinas county;
* Pregnant or lactating women;
* Patients with severe, non-stabilized neurological or psychiatric problems;
* Use of anti-obesity or lipid-lowering medication;
* Use of adrenergic or benzodiazepine drugs;
* Use of illicit drugs;
* Individuals with neoplasms, transmissible diseases, rheumatic disease, hepatic or renal insufficiency, non-treated thyroid dysfunction, diabetes mellitus, cardiovascular disease, history of fainting, active infection;
* Individuals who are allergic to nuts, soybean, oats, sesame or celery;
* Individuals who have had a change of more than 5% of their body weight in the last six months;
* Individuals who are carrying some kind of diet or modification to their habitual eating habits.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Activation of beige/brown adipose tissue - Volume | Three months
  Changes from baseline maximum Standardized Uptake Values (SUVmax) and mean Standardized Uptake Values (SUVmean), as assessed by PET/CT (FDG-18).
Activation of beige/brown adipose tissue - Temperature | Three months
  Changes from baseline BAT temperature, as assessed by Thermal Imaging.
Activation of beige/brown adipose tissue - Adipokines | Three months
  Changes from baseline BAT adipokines, as assessed by ELISA.
Activation of beige/brown adipose tissue - Activation Genes | Three months
  Changes from baseline BAT activation genes, as assessed by PCR.

SECONDARY OUTCOMES:
Basal metabolic rates (BMR) | Three months
  Changes from baseline BMR, as assessed by Indirect Calorimetry.
Metabolic markers | Three months
  Changes from baseline LDL, HDL, total cholesterol, triglycerides and glucose levels (mg/dL).
Hormones | Three months
  Changes from baseline insulin and leptin levels, as assessed by ELISA.
Inflammatory markers | Three months
  Changes from baseline inflammatory cytokines (TNF-α, IL1β, MCP1, IL-6 and IL-10), as assessed by ELISA.
Insulin Sensitivity | Three months
  Changes from baseline insulin sensitivity, as assessed by OGIS (insulin and glucose levels will be combined to report insulin sensitivity in ml minˆ-1 mˆ-2).

CONTACTS AND LOCATIONS:
Overall Officials: Marcela R Simoes, MS Candidate, Principal Investigator — University of Campinas; Licio A Velloso, Professor, Study Director — University of Campinas
Locations (1):
- School of Medical Sciences - University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Carpentier AC, Blondin DP, Virtanen KA, Richard D, Haman F, Turcotte EE. Brown Adipose Tissue Energy Metabolism in Humans. Front Endocrinol (Lausanne). 2018 Aug 7;9:447. doi: 10.3389/fendo.2018.00447. eCollection 2018. PMID 30131768
- [Background] Leitner BP, Huang S, Brychta RJ, Duckworth CJ, Baskin AS, McGehee S, Tal I, Dieckmann W, Gupta G, Kolodny GM, Pacak K, Herscovitch P, Cypess AM, Chen KY. Mapping of human brown adipose tissue in lean and obese young men. Proc Natl Acad Sci U S A. 2017 Aug 8;114(32):8649-8654. doi: 10.1073/pnas.1705287114. Epub 2017 Jul 24. PMID 28739898
- [Background] Rachid B, van de Sande-Lee S, Rodovalho S, Folli F, Beltramini GC, Morari J, Amorim BJ, Pedro T, Ramalho AF, Bombassaro B, Tincani AJ, Chaim E, Pareja JC, Geloneze B, Ramos CD, Cendes F, Saad MJ, Velloso LA. Distinct regulation of hypothalamic and brown/beige adipose tissue activities in human obesity. Int J Obes (Lond). 2015 Oct;39(10):1515-22. doi: 10.1038/ijo.2015.94. Epub 2015 May 21. PMID 25994805
- See also: ProLon, a Fasting Mimicking Diet — https://prolonfmd.com/